CLINICAL TRIAL: NCT01761266
Title: A Multicenter, Randomized, Open-Label, Phase 3 Trial to Compare the Efficacy and Safety of Lenvatinib (E7080) Versus Sorafenib in First-Line Treatment of Subjects With Unresectable Hepatocellular Carcinoma
Brief Title: A Multicenter, Open-Label, Phase 3 Trial to Compare the Efficacy and Safety of Lenvatinib (E7080) Versus Sorafenib in First-line Treatment of Participants With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-304; 2012-002992-33 (EudraCT Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; Neoplasms; Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — lenvatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenvatinib (Active Comparator): Participants received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the participant's body weight less than (<) 60 kg at baseline, orally, once daily (QD) in continuous 28-day treatment cycles up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Lenvatinib
- Sorafenib (Active Comparator): Participants received sorafenib 400 mg tablets, orally, twice daily (BID) in continuous 28-day treatment cycles up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
  Other Names: E7080, Lenvima
  Arms: Lenvatinib
Drug: Sorafenib — 400 mg twice daily (BID) oral dosing.
  Arms: Sorafenib

SUMMARY:
E7080-G000-304 is a multicenter, randomized, open-label, noninferiority Phase 3 study to compare the efficacy and safety of lenvatinib versus sorafenib as a first-line systemic treatment in participants with unresectable Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
1. Participants must have confirmed diagnosis of unresectable HCC with any of the following criteria:

   * Histologically or cytologically confirmed diagnosis of HCC.
   * Clinically confirmed diagnosis of HCC according to American Association for the Study of Liver Diseases (AASLD) criteria, including cirrhosis of any etiology or with chronic hepatitis B or C infection criteria
2. At least one measurable target lesion according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) meeting the following criteria:

   • Hepatic lesion
   1. The lesion can be accurately measured in at least one dimension as >=1.0 centimeter (cm) (viable tumor for typical; and longest diameter for atypical), and
   2. The lesion is suitable for repeat measurement.

      • Nonhepatic lesion
   3. Lymph node (LN) lesion that measures at least one dimension as >=1.5 cm in the short axis, except for porta hepatis LN that measures >=2.0 cm in the short axis.
   4. Non-nodal lesion that measures >=1.0 cm in the longest diameter Lesions previously treated with radiotherapy or locoregional therapy must show radiographic evidence of disease progression to be deemed a target lesion.
3. Participants categorized to stage B (not applicable for transarterial chemoembolization [TACE]) or stage C based on Barcelona Clinic Liver Cancer (BCLC) staging system.
4. Adequate bone marrow function, defined as:

   * Absolute neutrophil count (ANC) >=1.5 X 10^9 per liter (/L)
   * Hemoglobin (Hb) >=8.5 gram per deciliter (g/dL)
   * Platelet count >=75 X 10^9/L.
5. Adequate liver function, defined as:

   * Albumin >=2.8 g/dL
   * Bilirubin less than or equal to (<=) 3.0 mg/dL
   * Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine aminotransferase (ALT) <=5 X the upper limit of normal (ULN).
6. Adequate blood coagulation function, defined as international normalized ratio (INR) <=2.3.
7. Adequate renal function defined as creatinine clearance greater than (>) 40 milliliter per minute (mL/min) calculated per the Cockcroft and Gault formula.
8. Adequate pancreatic function, defined as amylase and lipase <=1.5 X ULN.
9. Adequately controlled blood pressure (BP) with up to 3 antihypertensive agents, defined as BP <=150/90 millimeters of mercury (mmHg) at Screening and no change in antihypertensive therapy within 1 week prior to the Cycle1/Day1.
10. Child-Pugh score A.
11. Eastern Cooperative Oncology Group (ECOG)- performance status (PS) 0 or 1.
12. Males or females aged at least 18 years (or any age >18 years as determined by country legislation) at the time of informed consent.
13. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 International Units Per Liter (IU/L) or equivalent units of BhCG).

    A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
14. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least 1 month before dosing).
15. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
16. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
17. Provide written informed consent.
18. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria

1. Imaging findings for HCC corresponding to any of the following:

   * HCC with >=50 percent liver occupation
   * Clear invasion into the bile duct
   * Portal vein invasion at the main portal branch (Vp4).
2. Participants who have received any systemic chemotherapy, including anti-vascular endothelial growth factor (VEGF) therapy, or any systemic investigational anticancer agents, including lenvatinib, for advanced/unresectable HCC. Note: Participants who have received local hepatic injection chemotherapy are eligible.
3. Participants who have received any anticancer therapy (including surgery, percutaneous ethanol injection, radio frequency ablation, transarterial [chemo] embolization, hepatic intra-arterial chemotherapy, biological, immunotherapy, hormonal, or radiotherapy) or any blood enhancing treatment (including blood transfusion, blood products, or agents that stimulate blood cell production, eg, granulocyte colony-stimulating factor [G-CSF]) within 28 days prior to randomization.
4. Participants who have not recovered from toxicities as a result of prior anticancer therapy, except alopecia and infertility. Recovery is defined as < Grade 2 severity per Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0).
5. Significant cardiovascular impairment: history of congestive heart failure > New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
6. Prolongation of corrected QT interval (QTc) interval to >480 millisecond (ms)
7. Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib in the opinion of the investigator.
8. Bleeding or thrombotic disorders or use of anticoagulants requiring therapeutic INR monitoring, eg, warfarin or similar agents. Treatment with low molecular weight heparin and factor X inhibitors which do not require INR monitoring is permitted. Antiplatelet agents are prohibited throughout the study.
9. Gastrointestinal bleeding event or active hemoptysis (bright red blood of at least 0.5 teaspoon) within 28 days prior to randomization.
10. Gastric or esophageal varices that require interventional treatment within 28 days prior to randomization. Prophylaxis with pharmacologic therapy (eg, nonselective beta-blocker) is permitted.
11. Active malignancy (except for HCC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 36 months.
12. Participants whose only target lesion(s) is in bone will be excluded.
13. Meningeal carcinomatosis.
14. Any history of or current brain or subdural metastases.
15. Participants having >1+ proteinuria on urine dipstick testing will undergo a 24-hour urine collection for quantitative assessment of proteinuria. Participants with a urine protein >=1g/24 hours will be ineligible.
16. Surgical arterial-portal venous shunt or arterial-venous shunt.
17. Any medical or other condition that in the opinion of the investigator would preclude the participant's participation in a clinical study.
18. Known intolerance to lenvatinib or sorafenib (or any of the excipients).
19. Human immunodeficiency virus (HIV) positive or active infection requiring treatment (except for hepatitis virus).
20. Any history of drug or alcohol dependency or abuse within the prior 6 months.
21. Any participant who cannot be evaluated by either triphasic liver computed tomography (CT) or triphasic liver Magnetic resonance imaging (MRI) because of allergy or other contraindication to both CT and MRI contrast agents.
22. Major surgery within 3 weeks prior to randomization or scheduled for surgery during the study.
23. Participants has had a liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2016-11-13 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (185):
- United States (21):
  - Facility # 1, Los Angeles, California
  - Facility # 1, Sacramento, California
  - Facility # 1, San Francisco, California
  - Facility # 1, Washington D.C., District of Columbia
  - Facility # 1, Tampa, Florida
  - Facility # 1, Duluth, Georgia
  - Facility # 1, Lawrenceville, Georgia
  - Facility # 1, Baltimore, Maryland
  - Facility # 1, Detroit, Michigan
  - Facility # 1, Kansas City, Missouri
  - Facility # 1, St Louis, Missouri
  - Facility # 1, East Orange, New Jersey
  - Facility # 1, Brooklyn, New York
  - Facility # 1, Lake Success, New York
  - Facility # 1, New York, New York
  - Facility # 1, Charlotte, North Carolina
  - Facility # 1, Durham, North Carolina
  - Facility # 1, Portland, Oregon
  - Facility # 1, Austin, Texas
  - Facility # 1, Lubbock, Texas
  - Facility # 1, Seattle, Washington
- Australia (7):
  - Facility # 1, Camperdown, New South Wales
  - Facility # 1, Wentworthville, New South Wales
  - Facility # 1, Woolloongabba, Queensland
  - Facility # 1, Fitzroy, Victoria
  - Facility # 1, Melbourne, Victoria
  - Facility # 2, Melbourne, Victoria
  - Facility # 1, Nedlands, Western Australia
- Belgium (3):
  - Facility # 1, Brussels
  - Facility # 1, Edegem
  - Facility # 1, Liège
- Facility # 1, Ottawa, Ontario, Canada
- China (21):
  - Facility # 1, Hefei, Anhui
  - Facility # 1, Beijing, Beijing Municipality
  - Facility # 2, Beijing, Beijing Municipality
  - Facility # 3, Beijing, Beijing Municipality
  - Facility # 1, Chongqing, Chongqing Municipality
  - Facility # 1, Fuzhou, Fujian
  - Facility # 2, Fuzhou, Fujian
  - Facility # 1, Guangzhou, Guangdong
  - Facility # 1, Harbin, Heilongjiang
  - Facility # 1, Changsha, Hunan
  - Facility # 1, Nanjing, Jiangsu
  - Facility # 1, Suzhou, Jiangsu
  - Facility # 1, Changchun, Jilin
  - Facility # 1, Dalian, Liaoning
  - Facility # 1, Jinan, Shandong
  - Facility # 1, Shanghai, Shanghai Municipality
  - Facility # 3, Shanghai, Shanghai Municipality
  - Facility # 1, Xi’an, Shanxi
  - Facility # 2, Xi’an, Shanxi
  - Facility # 1, Hangzhou, Zhejiang
  - Facility # 1, Tianjin, Zhejiang
- France (14):
  - Facility # 1, Nice, Alpes Maritimes
  - Facility # 1, Pessac, Gironde
  - Facility # 1, Toulouse, Haute Garonne
  - Facility # 1, Montpellier, Herault
  - Facility # 1, Rennes, Ille Et Vilaine
  - Facility # 1, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Facility # 1, Amiens, Somme
  - Facility # 1, Créteil, Val De Marne
  - Facility # 1, Bordeaux
  - Facility # 1, Lille
  - Facility # 1, Lyon
  - Facility # 1, Nord
  - Facility # 1, Paris
  - Facility # 1, Rhone
- Germany (7):
  - Facility # 1, Heidelberg, Baden-Wurttemberg
  - Facility # 1, Tübingen, Baden-Wurttemberg
  - Facility # 1, Marburg, Hesse
  - Facility # 1, Hanover, Lower Saxony
  - Facility # 1, Cologne, North Rhine-Westphalia
  - Facility # 1, Essen, North Rhine-Westphalia
  - Facility # 1, Mainz, Rhineland-Palatinate
- Hong Kong (4):
  - Facility # 1, Hong Kong
  - Facility # 2, Hong Kong
  - Facility # 3, Hong Kong
  - Facility # 1, Kowloon
- Facility # 1, Petah Tikva, Israel
- Italy (8):
  - Facility # 1, Torrette, Ancona
  - Facility # 1, Bari
  - Facility # 1, Benevento
  - Facility # 1, Bologna
  - Facility # 1, Napoli
  - Facility # 2, Napoli
  - Facility # 1, Palermo
  - Facility # 1, Roma
- Japan (25):
  - Facility # 1, Nagoya, Aichi-ken
  - Facility # 1, Kashiwa, Chiba
  - Facility # 1, Matsuyama, Ehime
  - Facility # 1, Kurume, Fukuoka
  - Facility # 1, Sapporo, Hokkaido
  - Facility # 2, Sapporo, Hokkaido
  - Facility # 1, Nishinomiya, Hyōgo
  - Facility # 1, Kanazawa, Ishikawa-ken
  - Facility # 1, Kawasaki, Kanagawa
  - Facility # 1, Yokohama, Kanagawa
  - Facility # 1, Tsu, Mie-ken
  - Facility # 1, Ōmura, Nagasaki
  - Facility # 1, Ōsaka-sayama, Osaka
  - Facility # 1, Bunkyo-Ku, Tokyo
  - Facility # 1, Chuo-ku, Tokyo
  - Facility # 1, Koto-ku, Tokyo
  - Facility # 1, Minato-ku, Tokyo
  - Facility # 1, Musashino, Tokyo
  - Facility # 1, Shimonoseki, Yamaguchi
  - Facility # 1, Fukuoka
  - Facility # 1, Hiroshima
  - Facility # 1, Okayama
  - Facility # 2, Osaka
  - Facility # 1, Saga
  - Facility # 2, Saga
- Malaysia (5):
  - Facility # 1, Kuantan, Pahang
  - Facility # 1, George Town, Pulau Pinang
  - Facility # 1, Miri, Sarawak
  - Facility # 1, Batu Caves, Selangor
  - Facility # 1, Kuala Lumpur
- Philippines (5):
  - Facility # 1, Cebu City
  - Facility # 2, Cebu City
  - Facility # 1, Davao City
  - Facility # 1, Quezon City
  - Facility # 2, Quezon City
- Poland (3):
  - Facility # 1, Gdansk
  - Facility # 1, Warsaw
  - Facility # 1, Wroclaw
- Russia (6):
  - Facility # 1, Arkhangelsk
  - Facility # 1, Moscow
  - Facility # 2, Moscow
  - Facility # 3, Saint Petersburg
  - Facility # 4, Saint Petersburg
  - Facility # 1, Ufa
- Singapore (4):
  - Facility # 1, Singapore
  - Facility # 2, Singapore
  - Facility # 3, Singapore
  - Facility # 4, Singapore
- South Korea (18):
  - Facility # 1, Goyang-si, Gyeonggi-do
  - Facility # 1, Seongnam-si, Gyeonggi-do
  - Facility # 2, Seongnam-si, Gyeonggi-do
  - Facility # 1, Suwon, Gyeonggi-do
  - Facility # 1, Daegu, Gyeongsangbuk-do
  - Facility # 1, Hwasun, Jeollanam-do
  - Facility # 1, Busan
  - Facility # 2, Busan
  - Facility # 3, Busan
  - Facility # 1, Incheon
  - Facility # 1, Seoul
  - Facility # 2, Seoul
  - Facility # 3, Seoul
  - Facility # 4, Seoul
  - Facility # 5, Seoul
  - Facility # 6, Seoul
  - Facility # 7, Seoul
  - Facility # 8, Seoul
- Spain (8):
  - Facility # 1, L'Hospitalet de Llobregat, Barcelona
  - Facility # 1, Santander, Cantabria
  - Facility # 1, Badajoz
  - Facility # 1, Girona
  - Facility # 1, Madrid
  - Facility # 2, Madrid
  - Facility # 3, Madrid
  - Facility # 4, Madrid
- Taiwan (12):
  - Facility # 1, Kaohsiung City
  - Facility # 2, Kaohsiung City
  - Facility # 1, Taichung
  - Facility # 2, Taichung
  - Facility # 1, Tainan
  - Facility # 2, Tainan
  - Facility # 1, Taipei
  - Facility # 2, Taipei
  - Facility # 3, Taipei
  - Facility # 4, Taipei
  - Facility # 5, Taipei
  - Facility # 1, Taoyuan
- Thailand (5):
  - Facility # 1, Bangkoknoi, Bangkok
  - Facility # 1, Pathum Wan, Bangkok
  - Facility # 1, Ratchathewi, Bangkok
  - Facility # 1, Muang, Changwat Chiang Rai
  - Facility # 1, Muang, Chiang Mai
- United Kingdom (7):
  - Facility # 2, London, Greater London
  - Facility # 1, London, Greater London
  - Facility # 3, London, Greater London
  - Facility # 1, Manchester, Greater Manchester
  - Facility # 1, Liverpool, Merseyside
  - Facility # 1, Glasgow, Strathclyde
  - Facility # 1, Birmingham, West Midlands

REFERENCES:
- [Derived] Piscaglia F, Ikeda K, Cheng AL, Kudo M, Ikeda M, Breder V, Ryoo BY, Mody K, Ren M, Ramji Z, Sung MW. Association between treatment-emergent hypertension and survival with lenvatinib treatment for patients with hepatocellular carcinoma in the REFLECT study. Cancer. 2024 Apr 15;130(8):1281-1291. doi: 10.1002/cncr.35185. Epub 2024 Jan 23. PMID 38261521
- [Derived] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Cheng AL, Vogel A, Tovoli F, Ueshima K, Aikata H, Lopez CL, Pracht M, Meng Z, Daniele B, Park JW, Palmer D, Tamai T, Saito K, Dutcus CE, Lencioni R. Overall survival and objective response in advanced unresectable hepatocellular carcinoma: A subanalysis of the REFLECT study. J Hepatol. 2023 Jan;78(1):133-141. doi: 10.1016/j.jhep.2022.09.006. Epub 2022 Sep 20. PMID 36341767
- [Derived] Huynh J, Cho MT, Kim EJ, Ren M, Ramji Z, Vogel A. Lenvatinib in patients with unresectable hepatocellular carcinoma who progressed to Child-Pugh B liver function. Ther Adv Med Oncol. 2022 Aug 24;14:17588359221116608. doi: 10.1177/17588359221116608. eCollection 2022. PMID 36051472
- [Derived] Vogel A, Qin S, Kudo M, Su Y, Hudgens S, Yamashita T, Yoon JH, Fartoux L, Simon K, Lopez C, Sung M, Mody K, Ohtsuka T, Tamai T, Bennett L, Meier G, Breder V. Lenvatinib versus sorafenib for first-line treatment of unresectable hepatocellular carcinoma: patient-reported outcomes from a randomised, open-label, non-inferiority, phase 3 trial. Lancet Gastroenterol Hepatol. 2021 Aug;6(8):649-658. doi: 10.1016/S2468-1253(21)00110-2. Epub 2021 Jun 2. PMID 34087115
- [Derived] Okusaka T, Ikeda K, Kudo M, Finn R, Qin S, Han KH, Cheng AL, Piscaglia F, Kobayashi M, Sung M, Chen M, Wyrwicz L, Yoon JH, Ren Z, Mody K, Dutcus C, Tamai T, Ren M, Hayato S, Kumada H. Safety and efficacy of lenvatinib by starting dose based on body weight in patients with unresectable hepatocellular carcinoma in REFLECT. J Gastroenterol. 2021 Jun;56(6):570-580. doi: 10.1007/s00535-021-01785-0. Epub 2021 May 4. PMID 33948712
- [Derived] Briggs A, Daniele B, Dick K, Evans TRJ, Galle PR, Hubner RA, Lopez C, Siebert U, Tremblay G. Covariate-adjusted analysis of the Phase 3 REFLECT study of lenvatinib versus sorafenib in the treatment of unresectable hepatocellular carcinoma. Br J Cancer. 2020 Jun;122(12):1754-1759. doi: 10.1038/s41416-020-0817-7. Epub 2020 Apr 8. PMID 32265508
- [Derived] Yamashita T, Kudo M, Ikeda K, Izumi N, Tateishi R, Ikeda M, Aikata H, Kawaguchi Y, Wada Y, Numata K, Inaba Y, Kuromatsu R, Kobayashi M, Okusaka T, Tamai T, Kitamura C, Saito K, Haruna K, Okita K, Kumada H. REFLECT-a phase 3 trial comparing efficacy and safety of lenvatinib to sorafenib for the treatment of unresectable hepatocellular carcinoma: an analysis of Japanese subset. J Gastroenterol. 2020 Jan;55(1):113-122. doi: 10.1007/s00535-019-01642-1. Epub 2019 Nov 12. PMID 31720835
- [Derived] Evans TRJ, Kudo M, Finn RS, Han KH, Cheng AL, Ikeda M, Kraljevic S, Ren M, Dutcus CE, Piscaglia F, Sung MW. Urine protein:creatinine ratio vs 24-hour urine protein for proteinuria management: analysis from the phase 3 REFLECT study of lenvatinib vs sorafenib in hepatocellular carcinoma. Br J Cancer. 2019 Jul;121(3):218-221. doi: 10.1038/s41416-019-0506-6. Epub 2019 Jun 28. PMID 31249394
- [Derived] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 154 investigative sites in Australia, Belgium, Canada, China, France, Germany, Hong Kong, Israel, Italy, Japan, South Korea, Malaysia, Philippines, Poland, Russia, Singapore, Spain, Taiwan, Thailand, United Kingdom, and the United States from 1 March 2013 to 10 March 2021.
Pre-assignment Details: A total of 1,492 participants were screened, 954 participants were enrolled and randomized, out of which 951 participants were treated in the study.
Period: Overall Study
Arm/Group | Lenvatinib | Sorafenib
Started | 478 | 476
Treated | 476 | 475
Completed | 0 | 0
Not Completed | 478 | 476
Not completed — Death | 415 | 402
Not completed — Lost to Follow-up | 8 | 12
Not completed — Withdrawal by Subject | 14 | 10
Not completed — Sponsor Decision | 41 | 52

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized.
Groups:
- Lenvatinib: Participants received lenvatinib capsules 12 mg based on the participant's body weight >=60 kg or 8 mg based on the participant's body weight <60 kg at baseline, orally, once daily (QD) in continuous 28-day treatment cycles up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Lenvatinib | Sorafenib | Total
Number analyzed (Participants) | 478 | 476 | 954
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.69) | 61.2 (12.01) | 61.3 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 75 | 148
  Male | 405 | 401 | 806
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 17
  Not Hispanic or Latino | 472 | 465 | 937
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 334 | 326 | 660
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 6 | 13
  White | 135 | 141 | 276
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Time Frame: From date of randomization until date of death from any cause (approximately up to 3.8 years)
Population: The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
months | 13.6 (12.1) [12.1 to 14.9] | 12.3 (10.4) [10.4 to 13.9]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first. Disease progression was defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: From the date of randomization to the date of first documentation of disease progression, or date of death, whichever occurred first (approximately up to 3.8 years)
Population: The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Lenvatinib: Subjects received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the subject's body weight less than (<) 60 kg at baseline, orally, once daily (QD) in continuous 28-day treatment cycles up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
months | 7.4 (6.9) [6.9 to 8.8] | 3.7 (3.6) [3.6 to 4.6]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization to the date of first documentation of disease progression based on mRECIST. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: The time from the date of randomization to the date of first documentation of disease progression (approximately up to 3.8 years)
Population: The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
months | 8.9 (7.4) [7.4 to 9.2] | 3.7 (3.6) [3.6 to 5.4]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: as for outcome 2
Population: The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
percentage of participants | 24.1 (20.2) [20.2 to 27.9] | 9.2 (6.6) [6.6 to 11.8]

5. Secondary Outcome: Time to Clinically Meaningful Worsening of Health Related Quality of Life (HRQoL) Assessed Using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 included 30 questions comprising 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social) and 9 symptom scales (fatigue, pain, nausea/vomiting, dyspnoea, appetite loss, insomnia, constipation, diarrhea and financial difficulties) and a single global health and QOL status score. Most questions used a 4-point scale (1=Not at all to 4=Very much); 2 questions used a 7-point scale (1= Very poor to 7=Excellent). All domain scores were calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: Baseline up to Off-Treatment Visit (approximately up to 3.8 years)
Population: The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
months | 1.7 (1.05) [1.05 to 1.84] | 1.8 (1.05) [1.05 to 1.84]

6. Secondary Outcome: Time to Clinically Meaningful Worsening of HRQoL Assessed Using - EORTC QLQ- Hepatocellular Carcinoma Domain (HCC 18)
Description: The EORTC QLQ-HCC-18 was an 18-item questionnaire design used along with the 30-item EORTC QLQ-C30. EORTC QLQ-HCC 18 questionnaire included 8 symptom scales such as fatigue, jaundice, body image, nutrition, pain, fever, sex life and abdominal swelling. Each individual item ranges from 1 to 4, where 1 = "not at all" and 4 = "very much." All domain scores were calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represented a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represented a high QoL, but a high score for a symptom scale/item represented a high level of symptomatology/problem. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: Baseline up to Off-Treatment Visit (approximately up to 3.8 years)
Population: The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
months
  Fatigue | 1.9 (1.81) [1.81 to 1.97] | 1.8 (1.74) [1.74 to 1.87]
  Jaundice | 4.6 (3.72) [3.72 to 5.52] | 3.7 (2.86) [2.86 to 4.73]
  Body Image | 2.8 (2.73) [2.73 to 3.68] | 1.9 (1.84) [1.84 to 2.73]
  Nutrition | 4.1 (3.68) [3.68 to 5.52] | 2.8 (2.04) [2.04 to 3.06]
  Pain | 2.7 (1.97) [1.97 to 2.83] | 2.8 (2.73) [2.73 to 3.72]
  Fever | 5.5 (4.57) [4.57 to 6.51] | 3.7 (2.99) [2.99 to 5.52]
  Sex Life | 7.4 (5.46) [5.46 to 9.17] | 6.7 (4.60) [4.60 to 13.78]
  Abdominal swelling | 7.4 (5.52) [5.52 to 9.24] | 7.4 (5.46) [5.46 to 10.13]

7. Secondary Outcome: Time to Clinically Meaningful Worsening of HRQoL Assessed Using EuroQol Five Dimension Health Questionnaire (EQ-5D-3L)
Description: The EuroQol five dimension health questionnaire (EQ-5D-3L) assesses quality of life along 5 dimensions. Participants rate 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranges from 3-15 with "3" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions. EQ-5D-3L also included an EQ visual analogue scale (VAS) that ranges between 100 (best imaginable health) and 0 (worst imaginable health). Decrease from baseline in EQ-5D-3L signifies improvement. Total index EQ-5D-3L summary score was weighted with a range of -0.594 (worst) to 1.0 (best). EQ-5D-3L also included an EQ health utilities index (HUI) where 1.00 indicated perfect health while a score of 0.00 indicated death. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: Baseline up to Off-Treatment Visit (approximately up to 3.8 years)
Population: The FAS included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
months
  VAS | 2.8 (2.17) [2.17 to 3.65] | 1.9 (1.84) [1.84 to 2.33]
  HUI | 2.8 (1.97) [1.97 to 3.52] | 1.9 (1.84) [1.84 to 2.66]

8. Secondary Outcome: Area Under the Plasma Drug Concentration-time Curve (AUC) for Lenvatinib
Description: AUC was assessed on Cycle 1 Day 1, Cycle 2 Day 1 and Cycle 1 Day 15. Summarized data for all time points was reported. As planned, data for this secondary endpoint was collected and analyzed up to the primary completion date.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1: pre-dose, 0.5-4 and 6-10 hours post-dose; Cycle 1 Day 15: pre-dose, 2-12 hours post-dose (cycle length= 28 days)
Population: The pharmacokinetic (PK) analysis set included all participants who had received at least 1 dose of lenvatinib and had at least 1 quantifiable lenvatinib concentration.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Lenvatinib 8 mg: Participants received lenvatinib capsules 12 mg based on the participant's body weight >=60 kg or 8 mg based on the participant's body weight <60 kg at baseline, orally, once daily (QD) in continuous 28-day treatment cycles up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
- Lenvatinib 12 mg: Participants received lenvatinib 12 mg capsules based on the participant's body weight (>=60 kg) at Baseline, orally, once daily in continuous 28-day treatment cycles up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
Arm/Group | Lenvatinib 8 mg | Lenvatinib 12 mg
Number analyzed (Participants) | 150 | 318
nanogram*hour per milliliter (ng*h/mL) | 1969.6 (743.0) | 2120.9 (685.6)

9. Other Pre Specified Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR, or stable disease (SD). Best overall response of SD must have been >=7 weeks after randomization. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference the baseline sum of the diameters of target lesions. SD was when a case does not qualify for either PR or PD and was new non-target lesions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions. As planned, data for this pre-specified endpoint was collected and analyzed up to the primary completion date.
Time Frame: as for outcome 2
Population: The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
percentage of participants | 75.5 (71.7) [71.7 to 79.4] | 60.5 (56.1) [56.1 to 64.9]

10. Other Pre Specified Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with a best overall response of CR or PR or durable SD (duration of SD >=23 weeks after randomization). For participants whose best overall response (BOR) was SD, the duration of SD was defined as the time from the date of randomization to the first documented PD or death, whichever occurred first. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference the baseline sum of the diameters of target lesions. SD was when a case does not qualify for either PR or PD. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions. As planned, data for this pre-specified endpoint was collected and analyzed up to the primary completion date.
Time Frame: as for outcome 2
Population: The FAS included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 478 | 476
percentage of participants | 59.0 (54.6) [54.6 to 63.4] | 38.4 (34.1) [34.1 to 42.8]

11. Other Pre Specified Outcome: Percent Change From Baseline in Serum Biomarker
Description: The serum biomarkers analysed were angiopoietin-2 (ANG2), fibroblast growth factor 19 (FGF19), fibroblast growth factor 21 (FGF21), fibroblast growth factor 23 (FGF23) and vascular endothelial growth factor (VEGF) as blood serum biomarkers, and protein induced by vitamin K absence or antagonist-II (PIVKA-II) as a blood tumor marker in serum. As planned, data for this pre-specified endpoint was collected and analyzed up to the primary completion date.
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1, Cycle 8 Day 1, Cycle 9 Day 1 and at the Off-Treatment Visit (approximately up to 3.8 years)
Population: The pharmacodynamics (PD) analysis set included all participants who received at least 1 dose of study drug and had evaluable PD data. Here "n" was participants who were evaluable for the outcome measure at given time points.
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Lenvatinib | Sorafenib
Number analyzed (Participants) | 66 | 48
percent change
  ANG 2: Cycle 1 Day 15 | -28.1 (15.94) [lower limit 15.94] | 8.9 (23.96) [lower limit 23.96]
  ANG 2: Cycle 2 Day 1 | -28.8 (16.53) [lower limit 16.53] | -0.9 (24.06) [lower limit 24.06]
  ANG 2: Cycle 3 Day 1 | -32.2 (23.23) [lower limit 23.23] | 0.5 (26.62) [lower limit 26.62]
  ANG 2: Cycle 4 Day 1 | -35.6 (22.91) [lower limit 22.91] | -4.5 (20.05) [lower limit 20.05]
  ANG 2: Cycle 5 Day 1 | -38.9 (19.83) [lower limit 19.83] | 7.0 (23.25) [lower limit 23.25]
  ANG 2: Cycle 6 Day 1 | -36.7 (23.59) [lower limit 23.59] | -3.6 (24.82) [lower limit 24.82]
  ANG 2: Cycle 7 Day 1 | -41.4 (21.20) [lower limit 21.20] | 1.0 (32.83) [lower limit 32.83]
  ANG 2: Cycle 8 Day 1 | -40.2 (25.33) [lower limit 25.33] | -6.7 (31.26) [lower limit 31.26]
  ANG 2: Cycle 9 Day 1 | -39.6 (14.04) [lower limit 14.04] | -1.1 (29.68) [lower limit 29.68]
  ANG 2: Off-Treatment | 11.7 (99.13) [lower limit 99.13] | 16.8 (27.88) [lower limit 27.88]
  FGF19: Cycle 1 Day 15 | 75.0 (155.01) [lower limit 155.01] | 1.3 (83.65) [lower limit 83.65]
  FGF19: Cycle 2 Day 1 | 66.5 (134.26) [lower limit 134.26] | 36.6 (119.65) [lower limit 119.65]
  FGF19: Cycle 3 Day 1 | 86.9 (123.85) [lower limit 123.85] | 22.8 (70.58) [lower limit 70.58]
  FGF19: Cycle 4 Day 1 | 208.1 (602.11) [lower limit 602.11] | 46.8 (214.14) [lower limit 214.14]
  FGF19: Cycle 5 Day 1 | 152.8 (228.37) [lower limit 228.37] | -1.0 (40.36) [lower limit 40.36]
  FGF19: Cycle 6 Day 1 | 119.8 (203.81) [lower limit 203.81] | 26.9 (67.13) [lower limit 67.13]
  FGF19: Cycle 7 Day 1 | 64.4 (101.97) [lower limit 101.97] | -5.9 (57.39) [lower limit 57.39]
  FGF19: Cycle 8 Day 1 | 95.8 (135.31) [lower limit 135.31] | 53.9 (113.79) [lower limit 113.79]
  FGF19: Cycle 9 Day 1 | 159.3 (202.00) [lower limit 202.00] | 56.6 (109.46) [lower limit 109.46]
  FGF19: Off-Treatment | 140.1 (270.73) [lower limit 270.73] | 9.0 (64.17) [lower limit 64.17]
  FGF 21: Cycle 1 Day 15 | 22.0 (75.22) [lower limit 75.22] | 4.0 (43.14) [lower limit 43.14]
  FGF 21: Cycle 2 Day 1 | 15.7 (77.44) [lower limit 77.44] | 18.6 (57.18) [lower limit 57.18]
  FGF 21: Cycle 3 Day 1 | 38.3 (38.3) [lower limit 38.3] | 49.4 (76.43) [lower limit 76.43]
  FGF 21: Cycle 4 Day 1 | 42.9 (145.43) [lower limit 145.43] | 32.8 (70.63) [lower limit 70.63]
  FGF 21: Cycle 5 Day 1 | 41.0 (95.97) [lower limit 95.97] | 31.1 (43.15) [lower limit 43.15]
  FGF 21: Cycle 6 Day 1 | 52.6 (168.22) [lower limit 168.22] | 23.2 (40.90) [lower limit 40.90]
  FGF 21: Cycle 7 Day 1 | 63.4 (128.34) [lower limit 128.34] | 23.7 (53.84) [lower limit 53.84]
  FGF 21 : Cycle 8 Day1 | 38.3 (115.53) [lower limit 115.53] | 17.0 (68.51) [lower limit 68.51]
  FGF 21: Cycle 9 Day1 | 59.1 (108.39) [lower limit 108.39] | 68.9 (103.55) [lower limit 103.55]
  FGF 21: Off-Treatment | 141.4 (340.51) [lower limit 340.51] | 104.9 (183.28) [lower limit 183.28]
  FGF 23: Cycle 1 Day15 | 23.9 (49.01) [lower limit 49.01] | -16.3 (36.14) [lower limit 36.14]
  FGF 23: Cycle 2 Day 1 | 20.9 (56.91) [lower limit 56.91] | -6.2 (48.18) [lower limit 48.18]
  FGF 23: Cycle 3 Day 1 | 25.5 (45.27) [lower limit 45.27] | 17.3 (75.25) [lower limit 75.25]
  FGF 23: Cycle 4 Day 1 | 29.5 (48.38) [lower limit 48.38] | 14.2 (49.29) [lower limit 49.29]
  FGF 23: Cycle 5 Day 1 | 29.6 (63.69) [lower limit 63.69] | 1.0 (47.28) [lower limit 47.28]
  FGF 23: Cycle 6 Day 1 | 26.3 (54.57) [lower limit 54.57] | -10.6 (46.15) [lower limit 46.15]
  FGF 23: Cycle 7 Day 1 | 31.5 (57.44) [lower limit 57.44] | 0.7 (46.95) [lower limit 46.95]
  FGF 23: Cycle 8 Day 1 | 38.1 (67.35) [lower limit 67.35] | 2.8 (43.84) [lower limit 43.84]
  FGF 23: Cycle 9 Day 1 | 23.2 (62.58) [lower limit 62.58] | 0.5 (38.74) [lower limit 38.74]
  FGF 23: Off-Treatment | 17.8 (73.59) [lower limit 73.59] | 14.2 (47.11) [lower limit 47.11]
  PIVKA-II: Cycle 1 Day 15 | 80.0 (171.41) [lower limit 171.41] | 166.9 (256.04) [lower limit 256.04]
  PIVKA-II: Cycle 2 Day 1 | 169.7 (329.33) [lower limit 329.33] | 243.8 (416.82) [lower limit 416.82]
  PIVKA-II: Cycle 3 Day 1 | 252.4 (611.40) [lower limit 611.40] | 218.7 (281.45) [lower limit 281.45]
  PIVKA-II: Cycle 4 Day 1 | 371.7 (812.45) [lower limit 812.45] | 196.2 (348.80) [lower limit 348.80]
  PIVKA-II: Cycle 5 Day 1 | 628.2 (1752.64) [lower limit 1752.64] | 369.5 (766.59) [lower limit 766.59]
  PIVKA-II: Cycle 6 Day 1 | 648.7 (2746.41) [lower limit 2746.41] | 415.7 (554.27) [lower limit 554.27]
  PIVKA-II: Cycle 7 Day 1 | 184.8 (352.75) [lower limit 352.75] | 703.6 (1226.58) [lower limit 1226.58]
  PIVKA-II: Cycle 8 Day 1 | 277.8 (481.53) [lower limit 481.53] | 724.0 (1257.87) [lower limit 1257.87]
  PIVKA-II: Cycle 9 Day 1 | 318.8 (577.21) [lower limit 577.21] | 859.1 (1492.93) [lower limit 1492.93]
  PIVKA-II: Off-Treatment | 809.3 (1827.42) [lower limit 1827.42] | 272.5 (489.60) [lower limit 489.60]
  VEGF: Cycle 1 Day 15 | 157.5 (300.21) [lower limit 300.21] | 97.4 (118.43) [lower limit 118.43]
  VEGF: Cycle 2 Day 1 | 128.9 (333.85) [lower limit 333.85] | 94.0 (180.80) [lower limit 180.80]
  VEGF: Cycle 3 Day 1 | 97.7 (162.39) [lower limit 162.39] | 66.0 (124.58) [lower limit 124.58]
  VEGF: Cycle 4 Day 1 | 113.4 (231.19) [lower limit 231.19] | 76.1 (111.20) [lower limit 111.20]
  VEGF: Cycle 5 Day 1 | 132.4 (249.59) [lower limit 249.59] | 116.2 (215.57) [lower limit 215.57]
  VEGF: Cycle 6 Day 1 | 113.1 (219.36) [lower limit 219.36] | 130.9 (341.12) [lower limit 341.12]
  VEGF: Cycle 7 Day 1 | 133.1 (383.43) [lower limit 383.43] | 96.9 (173.77) [lower limit 173.77]
  VEGF: Cycle 8 Day 1 | 148.7 (349.58) [lower limit 349.58] | 181.1 (399.67) [lower limit 399.67]
  VEGF: Cycle 9 Day 1 | 129.6 (215.05) [lower limit 215.05] | 135.6 (267.61) [lower limit 267.61]
  VEGF: Off-Treatment | 127.1 (266.64) [lower limit 266.64] | 147.8 (304.31) [lower limit 304.31]

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events were collected from first dose of study drug (Baseline) up to 30 days after last dose of study drug (approximately up to 8 years)
Description: The safety analysis set included all participants who received at least 1 dose of study drug. All-cause mortality was reported for all participants randomized.
Arm/Group | Lenvatinib | Sorafenib
All-Cause Mortality (participants affected / at risk) | 415/478 | 402/476
Serious Adverse Events (participants affected / at risk) | 209/476 | 149/475
Other Adverse Events (participants affected / at risk) | 469/476 | 469/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib (N=476) | Sorafenib (N=475)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Heart valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 12 (15) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 7 (8) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 11 (11)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (7) | 2 (5)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (8) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (4)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (3) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 7 (7) | 4 (4)
Portal vein thrombosis (Hepatobiliary disorders) | 4 (6) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (6) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (4) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (7) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (2) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 5 (6)
Hepatic pain (Hepatobiliary disorders) | 1 (4) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 4 (4)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 5 (7)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Perihepatic abscess (Infections and infestations) | 1 (3) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (2)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 7 (8) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 14 (14)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 3 (4)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 21 (35) | 3 (4)
Cerebral haemorrhage (Nervous system disorders) | 3 (5) | 0 (0)
Coma hepatic (Nervous system disorders) | 3 (4) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (4) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0)
Diplegia (Nervous system disorders) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (5) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (3) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Necrotising bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 6 (12)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (5) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 5 (6)
General physical health deterioration (General disorders) | 5 (5) | 3 (4)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (2)
Death (General disorders) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (2)
Sudden death (General disorders) | 1 (1) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 14 (22) | 8 (11)
Sepsis (Infections and infestations) | 7 (11) | 3 (4)
Peritonitis bacterial (Infections and infestations) | 2 (3) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib (N=476) | Sorafenib (N=475)
Ascites (Gastrointestinal disorders) | 63 (82) | 39 (54)
Constipation (Gastrointestinal disorders) | 76 (95) | 52 (62)
Diarrhoea (Gastrointestinal disorders) | 186 (406) | 223 (448)
Dyspepsia (Gastrointestinal disorders) | 31 (40) | 18 (20)
Nausea (Gastrointestinal disorders) | 90 (131) | 71 (94)
Stomatitis (Gastrointestinal disorders) | 45 (67) | 56 (76)
Vomiting (Gastrointestinal disorders) | 75 (110) | 37 (65)
Alanine aminotransferase increased (Investigations) | 53 (86) | 51 (108)
Aspartate aminotransferase increased (Investigations) | 64 (128) | 80 (173)
Blood alkaline phosphatase increased (Investigations) | 32 (59) | 29 (40)
Blood bilirubin increased (Investigations) | 67 (141) | 63 (128)
Electrocardiogram QT prolonged (Investigations) | 33 (59) | 24 (62)
Gamma-glutamyltransferase increased (Investigations) | 37 (60) | 27 (41)
Neutrophil count decreased (Investigations) | 41 (101) | 13 (21)
Platelet count decreased (Investigations) | 87 (260) | 59 (127)
Weight decreased (Investigations) | 149 (290) | 108 (182)
White blood cell count decreased (Investigations) | 47 (115) | 25 (55)
Decreased appetite (Metabolism and nutrition disorders) | 162 (269) | 126 (165)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 43 (88) | 38 (56)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (52) | 20 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 48 (55) | 28 (30)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 47 (56) | 25 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (59) | 18 (32)
Headache (Nervous system disorders) | 45 (57) | 39 (48)
Insomnia (Psychiatric disorders) | 33 (38) | 28 (34)
Proteinuria (Renal and urinary disorders) | 117 (363) | 55 (125)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (54) | 37 (46)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 113 (134) | 57 (69)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 (35) | 15 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (41) | 35 (46)
Rash (Skin and subcutaneous tissue disorders) | 46 (59) | 77 (105)
Hypertension (Vascular disorders) | 200 (419) | 147 (269)
Anaemia (Blood and lymphatic system disorders) | 35 (55) | 43 (104)
Thrombocytopenia (Blood and lymphatic system disorders) | 33 (81) | 28 (90)
Hypothyroidism (Endocrine disorders) | 81 (104) | 8 (9)
Abdominal distension (Gastrointestinal disorders) | 39 (57) | 24 (27)
Abdominal pain (Gastrointestinal disorders) | 82 (136) | 83 (111)
Abdominal pain upper (Gastrointestinal disorders) | 58 (82) | 41 (59)
Asthenia (General disorders) | 53 (122) | 48 (84)
Fatigue (General disorders) | 141 (226) | 120 (170)
Oedema peripheral (General disorders) | 67 (107) | 33 (45)
Pyrexia (General disorders) | 63 (79) | 61 (74)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (16) | 120 (140)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 128 (236) | 246 (614)
Dry mouth (Gastrointestinal disorders) | 32 (38) | 8 (8)
Dizziness (Nervous system disorders) | 29 (33) | 16 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (39) | 17 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (14) | 26 (52)
Hepatic encephalopathy (Nervous system disorders) | 24 (37) | 6 (6)
Haematuria (Renal and urinary disorders) | 25 (34) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 23 (26) | 25 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No